CLINICAL TRIAL: NCT03713294
Title: Phase II Trial of Sequential Treatment of Multiple Myeloma With Antibody Therapy
Brief Title: Dexamethasone, Elotuzumab, and Pomalidomide in Treating Patients With Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1884; NCI-2018-02140 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1884 (Other: Mayo Clinic); 18-003574 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2024-11

CONDITIONS: Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; elotuzumab; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (dexamethasone, elotuzumab, pomalidomide) (Experimental): Patients receive dexamethasone IV on days 1, 8, 15, and 22 of cycles 1-2 and IV on day 1 and PO on days 8, 15, and 22 of subsequent cycles and elotuzumab IV on days 1, 8, 15, and 22 of cycles 1-2 and day 1 of subsequent cycles. Patients also receive pomalidomide PO on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Biological: Elotuzumab; Drug: Pomalidomide

INTERVENTIONS:
Drug: Dexamethasone — Given IV and PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Biological: Elotuzumab — Given IV
  Other Names: BMS-901608; Empliciti; HuLuc-63; HuLuc63; PDL-063; PDL063
Drug: Pomalidomide — Given PO
  Other Names: 4-Aminothalidomide; Actimid; CC-4047; Imnovid; Pomalyst

SUMMARY:
This phase II trial studies how well dexamethasone, elotuzumab, pomalidomide work in treating patients with multiple myeloma that has not responded to previous treatment. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as elotuzumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Pomalidomide may stop the growth of multiple myeloma by blocking the growth of new blood vessels necessary for tumor growth. Giving dexamethasone, elotuzumab, pomalidomide may work better in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the overall response rate (ORR) of utilizing elotuzumab, pomalidomide and dexamethasone in patients with disease refractory to daratumumab.

SECONDARY OBJECTIVES:

I. To determine percentage of patients achieving complete response (CR) with the elotuzumab combination.

II. To determine progression-free survival (PFS) for treatment with the elotuzumab combination.

III. To determine safety profile for treatment with the elotuzumab combination. IV. To determine the overall survival (OS) for patients receiving treatment with the elotuzumab combination.

OUTLINE:

Patients receive dexamethasone intravenously (IV) on days 1, 8, 15, and 22 of cycles 1-2 and IV on day 1 and orally (PO) on days 8, 15, and 22 of subsequent cycles and elotuzumab IV on days 1, 8, 15, and 22 of cycles 1-2 and day 1 of subsequent cycles. Patients also receive pomalidomide PO on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months until progressive disease, then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Pathologically confirmed diagnosis of multiple myeloma and noted to have progressive disease (International Myeloma Working Group [IMWG] criteria).
* At least one prior line of therapy.
* Disease refractory to daratumumab as defined by disease progression while on or =< 60 days of completing treatment with a daratumumab-containing regimen as part of any prior line of therapy.
* Measurable disease =< 14 days prior to registration.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1 or 2.
* Absolute neutrophil count (ANC) >= 1,000 cell/mm^3 without growth factor support (obtained =< 14 days prior to registration).
* Platelet >= 50,000 cells/mm^3 for patients who have bone marrow plasmacytosis < 50% or >= 30,000 cells/mm^3 for patients who have bone marrow plasmacytosis of >= 50% (obtained =< 14 days prior to registration).
* Total bilirubin =< 1.5 x upper limit of normal (ULN) unless due to Gilbert's syndrome, in which case the direct bilirubin must be =< 1.5 x ULN (obtained =< 14 days prior to registration).
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 3 x ULN (obtained =< 14 days prior to registration).
* Prothrombin time (PT)/international normalized ratio (INR)/activated partial thromboplastin time (aPTT) =< 1.5 x ULN OR if patient is receiving anticoagulant therapy and PT/INR or aPTT is within target range of therapy (obtained =< 14 days prior to registration).
* Calculated or measured creatinine clearance >= 30 ml/min (obtained =< 14 days prior to registration).
* Negative urine or serum pregnancy test done =< 14 days prior to registration, for persons of childbearing potential only.

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Provide written informed consent.
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study).
* Willing to follow the requirements of the (Revlimid/Pomalyst) Risk Evaluation and Mitigation Strategies (REMS) program.

Exclusion Criteria:

* Non-secretory multiple myeloma (MM) or known immunoglobulin light chain (AL) amyloidosis.
* Clinically significant active infection requiring intravenous antibiotics (=< 14 days prior to registration).
* >= Grade 3 neuropathy and/or POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy.

  * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial.
* Concurrent therapy considered investigational.

  * NOTE: Patients must not be planning to receive any radiation therapy (except localized radiation for palliative care that must be completed prior to starting Cycle 1, Day 1).
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women.
  * Nursing women (lactating females are eligible provided that they agree not to breast feed while taking lenalidomide).
  * Men or women of childbearing potential who are unwilling to employ adequate contraception.
* Other active malignancy =< 3 years prior to registration.

  * EXCEPTIONS:

    * Adequately treated basal cell or squamous cell skin cancer.
    * Any in situ cancer.
    * Adequately treated Stage I or II cancer from which the patient is currently in complete remission, or
  * NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer.
* Major surgery =< 4 weeks prior to registration.
* History of stroke/intracranial hemorrhage =< 6 months prior to registration.
* Clinically significant cardiac illness including New York Heart Association (NYHA) Class III or Class IV heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, or >= Grade 3 cardiac arrhythmias noted =< 14 days prior to registration.
* Currently active, clinically significant hepatic impairment Child-Pugh class B or C according to the Child Pugh classification.
* Exhibiting clinical signs of meningeal involvement of multiple myeloma.
* Known severe chronic obstructive pulmonary disease or asthma defined as forced expiratory volume (FEV1) in 1 second < 60% of expected.
* Prior exposure to elotuzumab.
* Prior history of disease refractory to pomalidomide.
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection.
  * Symptomatic congestive heart failure.
  * Unstable angina pectoris.
  * Cardiac arrhythmia.
  * Or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sikander Ailawadhi, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Patients receive dexamethasone IV on days 1, 8, 15, and 22 of cycles 1-2 and IV on day 1 and PO on days 8, 15, and 22 of subsequent cycles and elotuzumab IV on days 1, 8, 15, and 22 of cycles 1-2 and day 1 of subsequent cycles. Patients also receive pomalidomide PO on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 70 [42 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate (ORR) defined as a partial response (PR), very good partial response (VGPR), complete response (CR) or stringent CR (sCR). CR and sCR are defined in Outcome 2. VGPR requires: serum and urine M-protein detectable by immunofixation but not on electrophoresis OR >= 90% reduction in serum M-protein and urine M-protein <100 mg/24 h. If the only measurable disease is FLC, a >90% reduction in the difference between involved and uninvolved FLC levels. PR requires: if present at baseline, >= 50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >= 90% or to <200 mg/24hrs. If the only measurable disease is FLC, a ≥50% reduction in the difference between involved and uninvolved FLC levels. If the only measurable disease is BM, a ≥ 50% reduction in BM PCs (provided the baseline PCs was ≥ 30%). If present at baseline, ≥ 50% reduction in the size (SPD) of soft tissue plasmacytomas.
Time Frame: 3 years
Measure: Number; unit: proportion of participants
Arm/Group | Treatment
Number analyzed (Participants) | 37
proportion of participants | 0.35

2. Secondary Outcome: Percentage of Patients Achieving CR
Description: Will be estimated by the number of patients who achieve a sCR or CR divided by the total number of evaluable patients. Complete Response (CR) is defined by all of the following: negative immunofixation of serum and urine; disappearance of any soft tissue plasmacytoma; <5% PCs in bone marrow; and if the only measurable disease is Free Light Chain (FLC), a normal FLC ratio. Stringent Complete Response (sCR) is defined as CR plus normal FLC ratio and absence of clonal circulating plasma cells (PCs) immunohistochemistry or 2- to 4- color flow cytometry.
Time Frame: 3 years
Measure: Number; unit: percentage of patients who achieve CR
Arm/Group | Treatment
Number analyzed (Participants) | 37
percentage of patients who achieve CR | 0

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from registration to time of disease progression or death due to any cause.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 37
months | 3.7 [2.9 to 11.1]

4. Secondary Outcome: Count of Patients That Experienced a Grade 3 or Greater Adverse Events
Description: The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. The table of these events is located in the adverse events section of this report.
Time Frame: 37 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 37
Participants | 27

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from registration to death due to any cause.
Time Frame: 62 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment
Number analyzed (Participants) | 37
Months | 56.7 [27.2 to NA] — Not enough events occurred to determine upper limit.

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 37 months and mortality was collected over 62 months.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 18/37
Serious Adverse Events (participants affected / at risk) | 12/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=37)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Edema limbs (General disorders) | 1 (2)
Edema trunk (General disorders) | 1 (2)
Fatigue (General disorders) | 1 (1)
Endocarditis infective (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (2)
Uterine infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Investigations - Other, specify (Investigations) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=37)
Anemia (Blood and lymphatic system disorders) | 33 (264)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 2 (2)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Fatigue (General disorders) | 27 (247)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (8)
Lymphocyte count increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 26 (181)
Platelet count decreased (Investigations) | 27 (102)
White blood cell decreased (Investigations) | 8 (19)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT03713294/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT03713294/ICF_001.pdf